CLINICAL TRIAL: NCT02131974
Title: Ultrasound Confirmation of Endotracheal Tube Location Using a Saline Filled Cuff
Acronym: ET_Tube
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Other Study IDs: HSC-MS-13-0324
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Pediatric Endotracheal Intubation (no Specific Condition)
Keywords: intubation, pediatric, endotracheal, cuffed ETT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research study is to help determine if the cuff of an endotracheal tube ( ETT) ( also known as a breathing tube)can be seen by ultrasound and to determine if visualization of this tube corresponds with correct tube depth. You are being asked to participate because you will be undergoing a cardiac catherization procedure which will involve endotracheal intubation.

Ultrasound is a safe technology that your doctor could possibly use to see the breathing tube. Right now, x-rays, which come with their own risks, are being used for this purpose. We are trying to see if we can avoid using x-rays.

This is a local study with 1 location. The study will enroll a total of 71 people. There is no sponsor for this study.

DETAILED DESCRIPTION:
If you enter the study, in the cardiac catheterization lab, after the anesthesiologist has done his part (placed the breathing tube while you are asleep and obtained the x-ray), we will use the ultrasound to check the position of the breathing tube. To help us see the breathing tube better, we will put some fluid in the cuff ( the balloon at the tip of the breathing tube). The tube may be repositioned as needed based on the chest x-ray. The entire procedure is estimated to take no more than 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish-speaking patients
* Age 0-21 years
* Elective cardiac catheterization procedure
* Endotracheal intubation with a cuffed ETT

Exclusion Criteria:

* Abnormal neck/tracheal anatomy
* Emergent cardiac catherization procedure
* Endotracheal intubation with an uncuffed ETT
* Inability to consent

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients scheduled to undergo elective cardiac catherization procedures will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2014-10-10 (Actual); Study Completion 2014-10-10 (Actual)

PRIMARY OUTCOMES:
Reliability of Ultrasound | 10 minutes
  Determine the reliability of ultrasound in visualizing a saline-filled cuff of the ETT in pediatric patients.

SECONDARY OUTCOMES:
Reliability of visualizing the cuff in patients without initial visualized cuff | 10 minutes
  In patients without an initial visualized cuff, determine the reliability of ultrasound in visualizing the cuff after a single retraction of the tube (as deemed permissible by cinefluoroscopy).

OTHER OUTCOMES:
Visualization of saline filled cuff | 10 minutes
  Determine if visualization of a saline-filled cuff at the suprasternal notch corresponds with correct tube depth as determined by cinefluoroscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Sakles JC, Laurin EG, Rantapaa AA, Panacek EA. Airway management in the emergency department: a one-year study of 610 tracheal intubations. Ann Emerg Med. 1998 Mar;31(3):325-32. doi: 10.1016/s0196-0644(98)70342-7. PMID 9506489
- [Background] Gausche M, Lewis RJ, Stratton SJ, Haynes BE, Gunter CS, Goodrich SM, Poore PD, McCollough MD, Henderson DP, Pratt FD, Seidel JS. Effect of out-of-hospital pediatric endotracheal intubation on survival and neurological outcome: a controlled clinical trial. JAMA. 2000 Feb 9;283(6):783-90. doi: 10.1001/jama.283.6.783. PMID 10683058
- [Background] Vanden Hoek TL, Morrison LJ, Shuster M, Donnino M, Sinz E, Lavonas EJ, Jeejeebhoy FM, Gabrielli A. Part 12: cardiac arrest in special situations: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S829-61. doi: 10.1161/CIRCULATIONAHA.110.971069. No abstract available. PMID 20956228
- [Background] Li J. Capnography alone is imperfect for endotracheal tube placement confirmation during emergency intubation. J Emerg Med. 2001 Apr;20(3):223-9. doi: 10.1016/s0736-4679(00)00318-8. PMID 11267809
- [Background] Galicinao J, Bush AJ, Godambe SA. Use of bedside ultrasonography for endotracheal tube placement in pediatric patients: a feasibility study. Pediatrics. 2007 Dec;120(6):1297-303. doi: 10.1542/peds.2006-2959. PMID 18055679
- [Background] Drescher MJ, Conard FU, Schamban NE. Identification and description of esophageal intubation using ultrasound. Acad Emerg Med. 2000 Jun;7(6):722-5. doi: 10.1111/j.1553-2712.2000.tb02055.x. No abstract available. PMID 10905655
- [Background] Werner SL, Smith CE, Goldstein JR, Jones RA, Cydulka RK. Pilot study to evaluate the accuracy of ultrasonography in confirming endotracheal tube placement. Ann Emerg Med. 2007 Jan;49(1):75-80. doi: 10.1016/j.annemergmed.2006.07.004. Epub 2006 Oct 2. PMID 17014927
- [Background] Weaver B, Lyon M, Blaivas M. Confirmation of endotracheal tube placement after intubation using the ultrasound sliding lung sign. Acad Emerg Med. 2006 Mar;13(3):239-44. doi: 10.1197/j.aem.2005.08.014. Epub 2006 Feb 22. PMID 16495415
- [Background] Kerrey BT, Geis GL, Quinn AM, Hornung RW, Ruddy RM. A prospective comparison of diaphragmatic ultrasound and chest radiography to determine endotracheal tube position in a pediatric emergency department. Pediatrics. 2009 Jun;123(6):e1039-44. doi: 10.1542/peds.2008-2828. Epub 2009 May 4. PMID 19414520
- [Background] Raphael DT, Conard FU 3rd. Ultrasound confirmation of endotracheal tube placement. J Clin Ultrasound. 1987 Sep;15(7):459-62. doi: 10.1002/jcu.1870150706. PMID 3134447
- [Background] Uya A, Spear D, Patel K, Okada P, Sheeran P, McCreight A. Can novice sonographers accurately locate an endotracheal tube with a saline-filled cuff in a cadaver model? A pilot study. Acad Emerg Med. 2012 Mar;19(3):361-4. doi: 10.1111/j.1553-2712.2012.01306.x. PMID 22435870
- [Background] Matsuo K, Akata T, Yamaura K, Morikawa K, Kandabashi T, Ueda N, Tohyama K, Takahashi S. [Intraoperative monitoring of pressure within saline-filled, endotracheal tube cuff in adult patients undergoing CO2 laser laryngomicrosurgery]. Masui. 2002 May;51(5):482-8. Japanese. PMID 12058429